CLINICAL TRIAL: NCT04875507
Title: The Use of a Positive Psychology Intervention (PPI) to Promote the Psychological Well-being of Children Living in Poverty: a Feasibility Randomized Controlled Trial
Brief Title: PPI to Promote the Psychological Well-being of Children Living in Poverty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PPI_poverty
Record Dates: First submitted 2021-04-20; First posted 2021-05-06 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Adolescent Development
Keywords: Poverty; Positive Psychology; Depressive symptoms; Self-esteem; Quality of life
MeSH Terms: conditions — Depression | interventions — Psychology, Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive psychology (Active Comparator): The experimental group(n=60), who will receive a 1.5-hour workshop covering positive psychology techniques delivered by a qualified research assistant, in groups of less than 5 people.
  Interventions: Behavioral: Positive Psychology
- Control (No Intervention): The control group will receive no intervention.

INTERVENTIONS:
Behavioral: Positive Psychology — This intervention aim to examine the effectiveness of PPI in reducing depressive symptoms, enhancing self-esteem, and promoting quality of life among Chinese children who are living in poverty. Participants in the experimental group will receive a 1.5 hour workshop on 4 positive psychology techniques, including (1) gratitude visit/letters, (2) 3 good things, (3) you at your best, and (4) using signature strengths. A booster intervention will be given at 1-week follow-up.
  Arms: Positive psychology

SUMMARY:
Positive psychology interventions use positive psychology techniques to identify meaning and value in life events to raise positive feelings and emotions. Application of PPIs has steadily increased in clinical and non-clinical samples. However, that meta-analysis did not include any study in a Chinese population, and it remains unclear whether PPIs are applicable in the Hong Kong Chinese context.

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted. A convenience sample of 120 patients age 13 to 17 years with no cognitive and/or behavioral problem(s) will be recruited in secondary school around Kwai Chung Estate Participants will be randomized into experimental and control group. The experimental group, who will receive a 1.5-hour workshop covering positive psychology techniques delivered by a qualified research assistant, in groups of less than 5 people, and a booster intervention at 1 week. The control group will received no intervention. Data collection will be conducted at baseline, 1 week, 1month, 3months and 6 months for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age from 13-17
* Can read Chinese and speak Cantonese

Exclusion Criteria:

* with identified cognitive and/or behavioral problem(s)
* with identified mental problem(s)
* participating in any mental health service/programme and/or receiving any psychiatric medication.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Screening rate | At baseline
  The number of children screened by the RA divided by the number of children available for screening during the recruitment period.
Eligibility rate | At baseline
  The number of eligible children divided by the number of screened children
Consent rate | At baseline
  The number of eligible children who consent to participate divided by the number of eligible children
Randomization rate | At baseline
  The number of children randomized to the experimental and control groups divided by the number of consenting children
Intervention attendance rate | Immediately after the training workshop
  The number of participants in the experimental group who complete the intervention divided by the number of participants randomized into the group
Intervention attendance rate at 1-week follow-up | At 1-week follow-up
  The number of participants in the experimental group who complete the intervention divided by the number of participants randomized into the group
Adherence to the intervention protocol at 1-week follow-up | At 1-week follow-up
  The number of participants in the experimental group who practice the skills gained divided by the number of participants randomized into the group
Retention rate at 6-month follow-up | At 6-month follow-up
  The number of participants who remain in this study divided by the number of randomized participants, calculated by group at each follow-up
Completion rate at 6-month follow-up | At 6-month follow-up
  The number of participants who return the questionnaires divided by the number of questionnaires distributed
Missing data at baseline | At baseline
  The percentage of missing in the dataset
Missing data at 1-week follow-up | At 1-week follow-up
  The percentage of missing in the dataset
Missing data at 1-month follow-up | At 1-month follow-up
  The percentage of missing in the dataset
Missing data at 3-month follow-up | At 3-month follow-up
  The percentage of missing in the dataset
Missing data at 6-month follow-up | At 6-month follow-up
  The percentage of missing in the dataset
Adverse events at baseline | At baseline
  unfavorable and unintended events
Adverse events at 1-week follow-up | At 1-week follow-up
  unfavorable and unintended events
Adverse events at 1-month follow-up | At 1-month follow-up
  unfavorable and unintended events
Adverse events at 3-month follow-up | At 3-month follow-up
  unfavorable and unintended events
Adverse events at 6-month follow-up | At 6-month follow-up
  unfavorable and unintended events

SECONDARY OUTCOMES:
Chinese version of the Rosenberg Self-esteem Scale at 6-month follow-up | At 6-month follow-up
  Assess participants' self-esteem
Chinese version of the Pediatric Quality of Life Inventory at 6-month follow-up | At 6-month follow-up
  Assess participants' quality of life
Chinese version of The Center for Epidemiologic Studies Depression Scale for Children at 6-month follow-up | At 6-month follow-up
  Assess participants' depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Ka Yan Ho, Hong Kong, Hong Kong,China, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho KY, Lam KKW, Bressington DT, Lin J, Mak YW, Wu C, Li WHC. Use of a positive psychology intervention (PPI) to promote the psychological well-being of children living in poverty: study protocol for a feasibility randomised controlled trial. BMJ Open. 2022 Aug 17;12(8):e055506. doi: 10.1136/bmjopen-2021-055506. PMID 35977772